CLINICAL TRIAL: NCT05246891
Title: Rehabilitation Nursing Program in Otolaryngology
Status: Completed | Type: Observational
Sponsor: University of Évora (Other)
Collaborators: Instituto Portugues Oncologia de Lisboa Francisco Gentil (Other)
Responsible Party: Principal Investigator, José Manuel Afonso Moreira, Principal Investigator, University of Évora
Other Study IDs: University of Évora
Record Dates: First submitted 2022-02-06; First posted 2022-02-18 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Rehabilitation; Neck Cancer; Otorhinolaryngologic Neoplasms
Keywords: Maxillofacial Surgery; Head and neck cancer; Otolaryngology
MeSH Terms: conditions — Head and Neck Neoplasms; Otorhinolaryngologic Neoplasms | interventions — Rehabilitation Nursing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rehabilitation nursing intervention: Functional respiratory rehabilitation exercise plan. Motor exercise plan. Cardiorespiratory optimization. Early diagnosis of potential problems associated.
  Interventions: Other: rehabilitation nursing
- Rehabilitation nursing not intervention: General nursing care
  Interventions: Other: rehabilitation nursing

INTERVENTIONS:
Other: rehabilitation nursing — Functional respiratory rehabilitation and motor exercise plan.

SUMMARY:
The European Commission's current political guidelines demonstrate into a joint plan aimed at improving and controlling cancer disease. Head and neck cancer (HNC) are the sixth most common cancer worldwide. The surgery is one of the most effective treatments, however it significantly compromises the self-care and functional capacity of the patients, so the intervention the Rehabilitation Nurse (RN) is essential.

Objective: Compare the degree of dependence in discharge from patients undergoing HNC surgery with RN intervention versus general nursing care (not RN intervention). The specific objective is to analyze the role of confounders in the effect of the RN intervention on the patient dependence.

Seventy-nine patients with RN intervention who undergoing a different type of surgery (1-Neck dissection, 2-Total laryngectomy with neck dissection, 3-Pelviglossomandibulectomy with neck dissection and tracheotomy, 4-Pelviglossomandibulectomy with neck dissection, pectorals major flap and tracheotomy) and all patients who undergoing the same type of surgery without RN intervention (n=72).

DETAILED DESCRIPTION:
Seventy-nine patients with RN intervention who undergoing a different type of surgery (1-Neck dissection, 2-Total laryngectomy with neck dissection, 3-Pelviglossomandibulectomy with neck dissection and tracheotomy, 4-Pelviglossomandibulectomy with neck dissection, pectorals major flap and tracheotomy) and all patients who undergoing the same type of surgery without RN intervention (n=72). Differences between groups were calculated using non-parametric tests Chi-square for categorical variables and Mann-Whitney U for numeric variable. After correlation tests between variables, statistical analysis was carried out through Poisson regression to a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing a different type of surgery: 1-Neck dissection, 2-Total laryngectomy with neck dissection, 3-Pelviglossomandibulectomy with neck dissection and tracheotomy, 4-Pelviglossomandibulectomy with neck dissection, pectorals major flap and tracheotomy.

Exclusion Criteria:

* Participants will be excluded if not be possible access of the clinical information.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a Head and Neck surgery after diagnosis of cancer.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change is being assessed | 0 week - 4 weeks
  Self-care: Barthel Index (0 points-100 points)

SECONDARY OUTCOMES:
Impatient days | 0 week - 4 weeks
  Days of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: José JM Moreira, MSc, Principal Investigator — University of Évora
Locations (1):
- University of Évora, Evora, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahlberg A, Engstrom T, Nikolaidis P, Gunnarsson K, Johansson H, Sharp L, Laurell G. Early self-care rehabilitation of head and neck cancer patients. Acta Otolaryngol. 2011 May;131(5):552-61. doi: 10.3109/00016489.2010.532157. PMID 21492066
- [Background] Clarke P, Radford K, Coffey M, Stewart M. Speech and swallow rehabilitation in head and neck cancer: United Kingdom National Multidisciplinary Guidelines. J Laryngol Otol. 2016 May;130(S2):S176-S180. doi: 10.1017/S0022215116000608. PMID 27841134
- [Background] Davidson A, Williams J. Factors affecting quality of life in patients experiencing facial disfigurement due to surgery for head and neck cancer. Br J Nurs. 2019 Feb 14;28(3):180-184. doi: 10.12968/bjon.2019.28.3.180. PMID 30746969
- [Background] Sheikh A, Shallwani H, Ghaffar S. Postoperative shoulder function after different types of neck dissection in head and neck cancer. Ear Nose Throat J. 2014 Apr-May;93(4-5):E21-6. PMID 24817237